CLINICAL TRIAL: NCT05415787
Title: Evaluation of the Technical Feasibility of Testing Circulating Tumour DNA for Homologous Recombination Gene Variants in Metastatic Prostate Cancer.
Brief Title: Evaluation of the Technical Feasibility of Testing ct DNA for Homologous Recombination Gene Variants in Metastatic Prostate Cancer.
Acronym: PROMECI
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR220119 PROMECI
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Circulating Tumor DNA; Metastatic Prostate Cancer
Keywords: Prostate cancer; ctDNA; HR genes
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample and Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with metastatic prostate cancer
  Interventions: Other: Blood sample; Other: Urine sample

INTERVENTIONS:
Other: Blood sample — 2 tubes Cell free DNA are taken during a blood sample already planned in the patient's care.
Other: Urine sample — Urine sample is taken during the consultation carried out for the patient's care

SUMMARY:
Evaluation of technical feasibility for Homologous Recombination (HR) genes variants research on circulating tumor DNA (ctDNA) from plasma and urine of patients with a metastatic prostate cancer.

DETAILED DESCRIPTION:
The benefit of PARPi has been well established for ovarian (SOLO-1 study) and prostate cancer (PROFOUND study) with defects in the Homologous Recombination Repair (HRR) system due to BRCA1 or BRCA2 variants. Somatic variants in HRR genes are currently researched by Next Generation Sequencing (NGS). However, in metastatic prostate cancer, using formalin-fixed and paraffin-embedded (FFPE) samples, failure rate is around 30 % according to our retrospective datas, in agreement with the data of the PROFOUND study, highlighting a real pre-analytical matter when FFPE samples are used for NGS testing. Research of such alterations on circulating tumor DNA (ctDNA) extracted from plasma or urine could be a promising alternative test.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years
* Metastatic prostate cancer
* Archived tissue sample available for testing for somatic variants of HRR genes (including BRCA1/BRCA2)
* Free, informed and signed consent for research

Non inclusion criteria

* Refusal of blood and urine collection
* Patient cognitively incapable of signing consent to participate in this study
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Circulating plasma tumour DNA | Baseline
  search for somatic variants of HRR genes (including BRCA1/BRCA2)
Circulating urine tumour DNA | Baseline
  search for somatic variants of HRR genes (including BRCA1/BRCA2)
FFPE tissue | Baseline
  search for somatic variants of HRR genes (including BRCA1/BRCA2)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Tallegas, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided